CLINICAL TRIAL: NCT02321098
Title: Determination of Antifungal Activity of Loceryl Nail Lacquer 5% When Used Concomitantly With a Cosmetic Nail Varnish Compared to a Loceryl Nail Lacquer (NL) 5% Alone in Treatment of Toenail Distal Subungual Onychomycosis
Brief Title: Antifungal Activity of Loceryl Nail Lacquer in Combination With a Cosmetic Varnish
Acronym: COOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD.03.SPR.29106; 2013-000544-26 (EudraCT Number)
Record Dates: First submitted 2014-12-08; First posted 2014-12-22 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Foot Dermatoses
Keywords: Onychomycosis; antifungal
MeSH Terms: conditions — Foot Dermatoses; Onychomycosis

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Only 12 first weeks of treatment with Loceryl NL and/or Loceryl alone were investigator masked and randomized.
  15 months of treatment with Loceryl NL alone had an open study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigator blinded Loceryl NL+ Cosmetic varnish (Experimental): Loceryl NL+ Cosmetic varnish once/week for 12 weeks on right or left foot toenails
  Interventions: Drug: Loceryl NL + Cosmetic varnish; Drug: Loceryl NL 15 months
- Investigator blinded Loceryl NL alone (Experimental): Loceryl NL once/week for 12 weeks on right or left foot toenails
  Interventions: Drug: Loceryl NL 12 weeks; Drug: Loceryl NL 15 months

INTERVENTIONS:
Drug: Loceryl NL + Cosmetic varnish — Loceryl NL + Cosmetic varnish once/week for 12 weeks
  Arms: Investigator blinded Loceryl NL+ Cosmetic varnish
Drug: Loceryl NL 12 weeks — Loceryl NL once/week for 12 weeks
  Arms: Investigator blinded Loceryl NL alone
Drug: Loceryl NL 15 months — Loceryl once/week for additional 15 months

SUMMARY:
The main objective is to compare efficacy, in terms of antifungal activity of Loceryl Nail Lacquer associated with a Cosmetic Varnish and Loceryl Nail Lacquer alone, in the treatment of mild to moderate toenail Distal Subungual Onychomycosis.

The second objective of this study will be photographic follow-up of clinical improvement and cure after the initial treatment period of 12 weeks, for 15 additional months.

DETAILED DESCRIPTION:
Study center:

A total of 50 subjects were to be included in 1 site in Iceland.

Methodology:

* Group Loceryl Nail Lacquer+ Cosmetic Varnish:

  * Loceryl Nail Lacquer to be applied once weekly for 12 weeks on all affected toenails,
  * Cosmetic varnish to be applied once weekly for 12 weeks on all affected toenails and/or all toenails.
* Group Loceryl Nail Lacquer alone:

  - Loceryl Nail Lacquer to be applied once weekly for 12 weeks on all affected toenails.
* All eligible subejct with no clinical sign of clinical aggravation of Onychomycosis at week 12, could continue to apply Loceryl Nail Lacquer alone, once a week for 15 additional months (or less in case of complete cure).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a mild to moderate Distal Subungual Onychomycosis (DSO) on at least 1 great toenail chosen as a Target nail
* Subjects must have maximum of 50% of nail distal edge involved
* Subjects with positive mycological results (direct microscopy and culture) of the Target nail for dermatophytes or Yeast (including Candida) at Screening

Exclusion Criteria:

* Subjects with clinically important abnormal physical findings at the Screening/Baseline visit
* Subjects with Lichen planus, eczema, psoriasis, or other abnormalities of the nail unit
* Subjects with known immunodeficiencies, radiation therapy, immune suppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Principal Investigator, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 50 subjects included to treat their affected toenails with Loceryl NL with or without Cosmetic Varnish for 12 weeks, First Subject In (FSI) = 11 Feb 2014, Last Subject Out (LSO) = 31 Oct 2014
  29 subjects without aggravation of their disease treated their toenails with Loceryl NL 15 additional months: FSI = 03 Nov 2014, LSO = 21Jan 2016
Pre-assignment Details: At screening all subjects had a mycological sampling of one of the diseased great toenails. Only screened subjects with both positive mycological results (direct microscopy and culture) at Baseline are randomized into one of the two arms for 12 weeks.
Groups:
- Loceryl NL+ Cosmetic Varnish: Loceryl NL + Cosmetic varnish once/week for 12 weeks
- Loceryl NL 15 Months: Loceryl NL once/week for additional 15 months
Period: 12 Weeks Treament
Arm/Group | Loceryl NL+ Cosmetic Varnish | Loceryl NL 12 Weeks | Loceryl NL 15 Months
Started | 26 | 24 | 0
Completed | 25 | 23 | 0
Not Completed | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Period: Additional 15 Months Treatment
Arm/Group | Loceryl NL+ Cosmetic Varnish | Loceryl NL 12 Weeks | Loceryl NL 15 Months
Started | 0 | 0 | 29
Completed | 0 | 0 | 21
Not Completed | 0 | 0 | 8
Not completed — Lack of Efficacy | 0 | 0 | 6
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Loceryl NL+Cosmetic Varnish: Loceryl NL+Cosmetic varnish once/week for 12 weeks
- Loceryl NL15 Months: Loceryl NL once/week for 15 months
- Total: Total of all reporting groups
Arm/Group | Loceryl NL+Cosmetic Varnish | Loceryl NL 12 Weeks | Loceryl NL15 Months | Total
Number analyzed (Participants) | 26 | 24 | 0 | 50
Age, Categorical [Count of Participants; unit: Participants] — Population: In Loceryl + cosmetic varnish arm 14 subjects out of 25 and 15 subjects out of 23 in Loceryl alone arm having completed 12 weeks Treatment period, continued to apply Loceryl for additional 15 months
  Participants
    Treatment period: <=18 years | 0 | 0 |  | 0
    Treatment period: Between 18 and 65 years | 18 | 18 |  | 36
    Treatment period: >=65 years | 8 | 6 |  | 14
Age, Continuous [Mean (Standard Deviation); unit: years] — Treatment period: 50 subjects are included in two arms for 12 weeks Population: From the 50 included subjects, 48 completed the study treatment period of 12 weeks and only 29 were eligible to continue to apply 15 additional months Loceryl NL
  years
    Treatment Period | 55.1 (12.0) | 53.7 (12.5) |  | 54.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Not all subjects randomized in treatment period (50) were eligible to apply Loceryl NL 15 additional months (29 subjects only were eligible)
  Participants
    Treatment Period: Female | 7 | 4 |  | 11
    Treatment Period: Male | 19 | 20 |  | 39
Region of Enrollment [Count of Participants; unit: Participants] — Population: In Loceryl + cosmetic varnish arm 14 subjects out of 25 and 15 subjects out of 23 in Loceryl alone arm having completed 12 weeks Treatment period, continued to apply Loceryl for additional 15 months
  Participants
    Iceland | 26 | 24 |  | 50

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Antifungal Activity of Loceryl Nail Lacquer
Description: Measurement of diameter of zones of inhibition (mm) produced by residual drug in toenails
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: Milimeter
Arm/Group | Loceryl NL+Cosmetic Varnish | Loceryl NL 12 Weeks
Number analyzed (Participants) | 25 | 23
Milimeter | 53.6 (9.1) | 53.5 (6.2)

2. Secondary Outcome: Absence of Dermatophytes in Nail Samples Culture
Time Frame: Week 12
Measure: Number; unit: participants
Groups:
- Loceryl NL+ Cosmetic Varnish + Loceryl NL: Once weekly application of Loceryl NL + Cosmetic varnish during 12 weeks followed by Loceryl NL once weekly applications for 15 additional months
- Loceryl NL + Loceryl NL: Once weekly application of Loceryl NL alone during 12 weeks followed by Loceryl NL once weekly applications for 15 additional months
Arm/Group | Loceryl NL+ Cosmetic Varnish + Loceryl NL | Loceryl NL + Loceryl NL
Number analyzed (Participants) | 25 | 23
participants | 25 | 23

ADVERSE EVENTS:
Time Frame: Adverse events are collected during both study periods (Treatment period of 12 weeks and additional period of 15 months treatment)
Groups:
- Loceryl NL 12 Weeks: Loceryl NL alone once/week for 12 weeks
Arm/Group | Loceryl NL+Cosmetic Varnish | Loceryl NL 12 Weeks | Loceryl NL 15 Months
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24 | 2/29
Other Adverse Events (participants affected / at risk) | 3/26 | 4/24 | 10/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loceryl NL+Cosmetic Varnish (N=26) | Loceryl NL 12 Weeks (N=24) | Loceryl NL 15 Months (N=29)
CARCINOMA SQUAMOCELLULARE IN LEFT TONSILLARY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loceryl NL+Cosmetic Varnish (N=26) | Loceryl NL 12 Weeks (N=24) | Loceryl NL 15 Months (N=29)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 3 (3) | 5 (8)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
TONSILLITIS (Infections and infestations) | 2 (2) | 0 (0) | 2 (3)
SINUSITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes